CLINICAL TRIAL: NCT02579837
Title: CLEAR SIGHT: A Randomized Trial of Non-Mydriatic Ultra-Widefield Retinal Imaging to Screen for Diabetic Eye Disease
Brief Title: CLEAR SIGHT: A Trial of Non-Mydriatic Ultra-Widefield Retinal Imaging to Screen for Diabetic Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Selina Liu, Assistant Professor, Division of Endocrinology & Metabolism, Department of Medicine, Schulich School of Medicine & Dentistry, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 106583
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy
Keywords: screening
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Screening (No Intervention): Participants randomized to the Usual Screening group will be advised by their Endocrinologist during their Diabetes Clinic visit to arrange an eye examination with their usual eye care professional (as per current standard of care).
- On-Site Screening (Experimental): Participants randomized to the On-Site Screening group will be advised by their Endocrinologist during their Diabetes Clinic visit to arrange an eye examination with their usual eye care professional (as per current standard of care). However, they will also undergo non-mydriatic ultra-widefield (UWF) retinal imaging (both 100 and 200 degrees) using the Optos 200Tx UWF retinal imaging device in the Ophthalmology Department on the same day as their Diabetes Clinic visit.
  Half of this group will by random allocation undergo optical coherence tomography (OCT) using the Zeiss Cirrus OCT, which may or may not be done on the same day (for practical reasons regarding availability of OCT at the hospital).
  Interventions: Device: Optos 200Tx; Device: Zeiss Cirrus

INTERVENTIONS:
Device: Optos 200Tx — non-mydriatic ultra-widefield (UWF) retinal imaging device
  Arms: On-Site Screening
Device: Zeiss Cirrus — optical coherence tomographer (OCT)
  Arms: On-Site Screening

SUMMARY:
Diabetic eye disease causes major vision loss in many Canadians and is costly. There are effective preventions and treatments for diabetic eye disease but they strongly depend upon regular screening in asymptomatic patients. The 2013 Canadian Diabetes Association (CDA) guidelines recommend annual screening by eye care professionals, either in-person or through interpretation of dilated pupil retinal photographs.

Despite the benefits of screening, adherence to these guidelines is poor. Reasons include patient barriers, i.e. need for eye drops, time off work, wait times, and transportation issues. An option to minimize these barriers is to screen using a camera called non-mydriatic ultra-widefield (UWF) retinal imaging. This can be quickly done without eye drops on the same day as patients' regularly scheduled diabetes clinic visits.

In this study, the investigators will compare the UWF camera to the usual screening approach recommended by the CDA. The investigators will invite 740 patients with diabetes due for eye screening to either be screened using the UWF camera on the day of their diabetes clinic visit or be screened by their usual eye care professional. The investigators' prediction is that same-day screening with UWF imaging will find more patients with diabetic eye disease who need treatment compared to usual screening.

DETAILED DESCRIPTION:
In this study, the investigators are addressing a significant and expanding "care-gap" question for patients with diabetes who are at risk for diabetic retinopathy (DR). DR is a major cause of impaired health-related quality of life in Ontarians through visual loss including blindness. Because the prevalence of DM in Ontario is increasing, the number of Ontarians over age 40 years with sight-threatening DR has been projected to increase by ~ 60% by 2031. DR is also a major source of health care costs: in 2007 the estimated health care system expenditure for vision loss from DR in Canada was $205 million.

There are proven effective strategies to prevent and treat DR. These strategies strongly depend upon regular screening in asymptomatic patients. Thus, the 2013 CDA practice guidelines recommended annual eye screening by experienced eye care professionals either in-person or through interpretation of dilated pupil retinal photographs and yet, despite the benefit of screening, adherence to the CDA guidelines is poor. At least part of this is due to patient-centered barriers including the need for mydriasis, time off of work, wait times, and transportation issues. Recent studies indicate that non-mydriatic UWF retinal imaging minimizes these barriers and also accurately detects clinically important DR as compared to reference standard tests (dilated pupil eye exam by an eye care professional or 7-field stereoscopic colour fundus photography).

In this study, the investigators' primary goal is to confirm or refute the hypothesis that screening by non-mydriatic UWF imaging at the time diabetes patients are seen for their routinely scheduled diabetes clinic visit (On-site Screening) improves the rate of detection of clinically important DR as compared to Usual Screening by the CDA guidelines. While the investigators are not testing the effect of screening by non-mydriatic UWF on visual outcomes, confirmation of the investigators' hypothesis has the potential to improve current screening strategies for DR in Ontario and, with that, an expectation that this will reduce vision-threatening diabetic eye disease.

ELIGIBILITY:
Inclusion Criteria:

1. Known diagnosis of Type 1 diabetes for >/= 5 years or Type 2 diabetes of any duration
2. At least 12 months since the last screening for diabetic eye disease by an eye care professional as this is based on patient self-report. Subsequent confirmation of the date of the last eye examination will be obtained via communication with the patient's eye care professional. Patients who indicate by self-report that it has been more than a year since screening, but in whom it is subsequently confirmed that their last screen occurred <12 months prior to entry, will be randomized but will not be included in the primary analysis comparing On-Site to Usual Screening.
3. Provision of informed consent

Exclusion Criteria:

1. Under active followup by an ophthalmologist for DM-related eye disease. Active followup requires that, at recruitment, the patient is scheduled for a future ophthalmologist appointment for any reason.
2. Inability to provide informed consent.
3. Any other condition or circumstance which in the judgment of the investigator makes it unlikely that the patient can adhere to the study protocol. This includes co-morbidities for which expected life-expectancy is less than a year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2016-03; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with Actionable Eye Disease (AED) | within 12 months of randomization
  Usual Screening Group: AED will be based upon DR grading and the disposition recommendation as that information is provided on the exam report from the participant's usual eye care professional. Any one of the following will be considered indicative of AED if noted on the report: a) moderate or severe non-proliferative DR; b) any proliferative DR; c) clinically significant macular edema (CSME); d) referral to an ophthalmologist; e) recommendation for re-examination in <12 months.
  On-Site Screening Group: AED will be based on interpretation of non-mydriatic UWF images by a retinal specialist where AED will require at least 1 finding of: DR (intra-retinal microvascular abnormalities or venous beading >/= 2 quadrants, neovascularization elsewhere, neovascularization of the disc, vitreous hemorrhage) or diabetic maculopathy (microaneurysms, retinal hemorrhages or exudates within 1 disc diameter of the fovea)

SECONDARY OUTCOMES:
Screening Adherence (rate of screening via primary assigned screening method) | within 12 months of randomization
  Determined by (i) the proportions of participants who have screening completed within 12 months of randomization by the primary screening method, viz., non-mydriatic UWF images (On-site Screening group) or an eye examination by an eye care professional (Usual Screening group); (ii) for participants in the On-site Screening group, the proportion who have also had a screening eye examination by an eye care professional within 1 year of randomization. For (i) and (ii) above, documentation of a screening examination by an eye care professional will require that the exam findings be provided in a written report
Proportion of participants with Diabetic Maculopathy (DME) | within 12 months of randomization
  Defined by: (i) the proportions of participants with clinically important macular edema detected by the primary screening method viz., non-mydriatic UWF images (On-site Screening group) or an eye examination by an eye care professional (Usual Screening group); (ii) the proportions of participants with DME detected by non-mydriatic UWF imaging alone versus non-mydriatic UWF imaging plus OCT; (iii) the proportions of participants with DME detected by non-mydriatic UWF imaging plus OCT versus eye examination by an eye care professional. The criteria to define DME by OCT are the presence of 1 or more of: intraretinal cysts, intraretinal exudates or subretinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Selina L Liu, MD MSc FRCPC, Principal Investigator — Western University
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu SL, Mahon LW, Klar NS, Schulz DC, Gonder JR, Hramiak IM, Mahon JL. A randomised trial of non-mydriatic ultra-wide field retinal imaging versus usual care to screen for diabetic eye disease: rationale and protocol for the Clearsight trial. BMJ Open. 2017 Aug 3;7(8):e015382. doi: 10.1136/bmjopen-2016-015382. PMID 28775182